CLINICAL TRIAL: NCT06939972
Title: A Single Group Study to Evaluate the Effects of a Topical Product on Cramps Associated With the Menstrual Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rael (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20674
Record Dates: First submitted 2025-01-05; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Dysmenorrhea; Menstrual Cramps
Keywords: Headaches; Mood changes; Fatigue
MeSH Terms: conditions — Dysmenorrhea; Headache; Fatigue | interventions — Analgesics; Camphor; Menthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical Product Application (Experimental): Participants will apply a topical product containing Camphor (4%) and Menthol (4%) to areas experiencing pain, such as the lower abdomen or lower back, during menstrual cycles.
  Interventions: Dietary Supplement: Topical Analgesic with Camphor and Menthol

INTERVENTIONS:
Dietary Supplement: Topical Analgesic with Camphor and Menthol — Participants will apply the product directly to the lower abdomen or back during menstrual cycles, following specific application instructions. The product provides analgesic and cooling effects to reduce discomfort.

SUMMARY:
This study evaluates the effectiveness of a topical product in reducing discomfort associated with menstrual cramps and back pain. Participants will apply the product during two menstrual cycles and complete study-specific questionnaires to assess the impact on symptoms and user perceptions.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-35.
* Has had a regular menstrual cycle for the past six months and is to predict their menstrual cycle and the timing of their menstruation.
* Mild to moderate self-reported discomfort during menstruation related to pelvic cramps and back pain.
* Generally healthy and not living with any uncontrolled chronic disease.
* Has a menstrual cycle between 21 and 35 days in length.
* Willing to maintain current diet, sleep, and activity level for the duration of the study.
* Resides in the United States.

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Current use of any blood thinning medication.
* Anyone with known severe allergic reactions.
* Anyone with any allergies requiring the use of an Epi-Pen.
* Anyone with any allergies or sensitivities to any of the study product ingredients.
* Anyone who is pregnant, breastfeeding, or trying to conceive currently or at any point until the end of the study period.
* Anyone unwilling to follow the study protocol.
* Anyone taking prescription medications for acute or chronic pain.
* Anyone with a diagnosis of a condition relating to the menstrual cycle or reproductive system-e.g., polycystic ovary syndrome (PCOS), premenstrual dysphoric disorder (PMDD), endometriosis, etc.
* Anyone diagnosed with other conditions that may cause lower back, abdominal, or pelvic discomfort- e.g., fibromyalgia, Crohn's, IBS, UC, chronic constipation, frequent UTIs, bacterial vaginosis (BV), or history or kidney stones.
* Anyone who has changed their birth control in the past three months.
* Anyone who has had any surgeries or invasive treatments in the past six months or has any planned up until the end of the study period.
* Anyone with any major illness in the past three months.
* Anyone currently experiencing symptoms associated with perimenopause.
* Anyone taking part in any other clinical trials or studies during this study's duration.
* Anyone with a history of substance abuse.
* Anyone who is currently a smoker or has been in the past three months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Reduction in Menstrual Cramps and Pain | Baseline, Day 5 of Cycle 1 (cycle 1 is 4 weeks), and Day 5 of Cycle 2 (cycle 2 is 4 weeks)
  Change in participant-reported menstrual cramps and associated pain severity, as assessed by a study-specific questionnaire.

SECONDARY OUTCOMES:
Participant Perception of Product Effectiveness | Baseline, Day 5 of Cycle 1 (cycle 1 is 4 weeks), and Day 5 of Cycle 2 (cycle 2 is 4 weeks)
  Evaluation of participants' perceptions of the product's effectiveness in alleviating menstrual cramps and symptoms, as assessed by a study-specific questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No